CLINICAL TRIAL: NCT02744547
Title: Effect of Spirulina on Serum Hyaluronic Acid as a Marker for Liver Fibrosis in Beta Thalassemic Children With Hepatitis C
Brief Title: Effect of Spirulina on Serum Hyaluronic Acid in Beta Thalassemic Children With Hepatitis C
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Tanta University (Other)
Responsible Party: Principal Investigator, Professor Mohamed Elshanshory, head of pediatric hematology and oncology unit, Tanta University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: 2900/11/14
Record Dates: First submitted 2016-04-16; First posted 2016-04-20 (Estimated); Last update posted 2019-04-10 (Actual); Status verified 2019-04

CONDITIONS: Beta Thalassemia Major
MeSH Terms: conditions — beta-Thalassemia

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- thalassemic children with hepatitis C (Experimental): 30 multitransfused beta thalassemic children infected with hepatitis C virus diagnosed by serological detection of HCV-antibodies and HCV RNA by polymerase chain reaction will be given Spirulina in a dose of 250 mg/kg/day orally for 3 months.
  Interventions: Dietary Supplement: Spirulina
- thalassemic children without hepatitis C (No Intervention): 30 multitransfused beta thalassemic children without hepatitis C virus infection

INTERVENTIONS:
Dietary Supplement: Spirulina — Spirulina in a dose of 250 mg/kg/day will be given orally for 3 months.
  Arms: thalassemic children with hepatitis C

SUMMARY:
Thalassemics can develop liver fibrosis because of iron overload and hepatitis C infection. The latter is the main risk factor for liver fibrosis in transfusion dependent thalassemics. Excess liver iron is clearly recognized as a co factor for the development of advanced fibrosis in patients with hepatitis virus C infection. Hyaluronic acid serum levels correlate with histological stages of liver fibrosis in hepatitis C patients, so it has a good diagnostic accuracy as a non invasive assessment of fibrosis and cirrhosis.there is evidence that suggests Spirulina may help to protect against liver damage, cirrhosis and liver failure in those with chronic liver disease.

ELIGIBILITY:
Inclusion Criteria:

* multitransfused beta thalassemic children with and without super added hepatitis C virus (HCV) infection diagnosed by serological detection of HCV antibodies and HCV RNA by polymerase chain reaction.

Exclusion Criteria:

* liver decompensation child younger than 3 years patients with hepatitis B infection

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Actual)
Dates: Start 2015-12 (Actual); Primary Completion 2017-12 (Actual); Study Completion 2017-12 (Actual)

PRIMARY OUTCOMES:
serum hyaluronic acid levels | 3 months

SECONDARY OUTCOMES:
liver function tests | 3 months
aspartate aminotransferase to platelet ratio index (APRI) | 3 months

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine- Tanta University, Tanta, Gharbia Governorate, Egypt